CLINICAL TRIAL: NCT05077072
Title: Opioid-Sparing Interdisciplinary Interventions Addressing Pain in Head and Neck Cancer Patients
Brief Title: Interdisciplinary Interventions to Address Pain Management Among Head and Neck Cancer Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0337; NCI-2021-09426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0337 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-22; First posted 2021-10-13 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Counseling; Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM I (CHAT) (Experimental): Patients participate in CHAT counseling intervention over 45-60 minutes twice a month for up to 12 weeks.
  Interventions: Other: Counseling; Other: Questionnaire Administration
- ARM II (NFB) (Experimental): Patients undergo NFB intervention over 20-30 minutes twice a week for up to 10 weeks.
  Interventions: Procedure: Electroencephalography; Behavioral: Neurofeedback; Other: Questionnaire Administration
- ARM III (SOC) (Active Comparator): Patients receive 2-3 standard of care sessions per month over 45-60 minutes for up to 12 weeks.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive SOC
  Other Names: standard of care; standard therapy
  Arms: ARM III (SOC)
Other: Counseling — Participate in CHAT counseling intervention
  Other Names: Counseling Intervention
  Arms: ARM I (CHAT)
Procedure: Electroencephalography — Undergo EEG
  Other Names: EEG; electroencephalogram
  Arms: ARM II (NFB)
Behavioral: Neurofeedback — Undergo NFB intervention
  Other Names: EEG biofeedback
  Arms: ARM II (NFB)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial compares different pain management interventions (standard of care [SOC], neurofeedback [NFB] training, and compassionate high alert team [CHAT]) in patients diagnosed with head and neck cancer who are at risk of developing non-medical opioid use (NMOU). The current standard treatment includes regular clinic visits and supportive care and counseling (including topics like patient-doctor communication, cancer care goals, financial issues counseling, and other topics). NFB training is a type of therapy that uses an electroencephalograph (EEG) and a computer software program to measure brain wave activity. The goal of NFB is to help teach patients with pain how to change their own brain waves to lower their feelings of pain and help improve their quality of life. CHAT is a supportive care intervention that includes symptom and pain management, counseling (about pain, symptoms, opioid use and safety, stress, and quality of life), and support for patients and their family members. NFB and CHAT may help to manage pain and lower patient use of opioids.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To test the hypothesis that this study will be feasible, as defined by adequate rates of adherence in the CHAT and NFB groups.

SECONDARY OBJECTIVES:

I. To examine the frequency of NMOU behaviors at the end of 3 months after CHAT, NFB, and SOC.

II. Examine the pain severity (area under the curve [AUC]), daily opioid use AUC of the cumulative morphine equivalent daily dose (MEDD), and mood (Hospital Anxiety and Depression Scale, HADS) for each of the treatment arms (CHAT, NFB, or SOC) in head and neck cancer (HNC) patients receiving radiation therapy at the end of 3 months.

EXPLORATORY OBJECTIVE:

I. To examine the cortical and subcortical regions of the brain associated with pain and our interventions (CHAT, NFB, and SOC) and the extent to which changes in electroencephalogram (EEG) patterns mediate the effects of the intervention.

OUTLINE: Patients are randomized into 1 of 3 arms.

ARM I: Patients participate in CHAT counseling intervention over 45-60 minutes twice a month for up to 12 weeks.

ARM II: Patients undergo NFB intervention over 20-30 minutes twice a week for up to 10 weeks.

ARM III: Patients receive 2-3 standard of care sessions per month over 45-60 minutes for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HNC, with patient scheduled to receive radiation therapy, with or without evidence of active disease
* Willingness to be seen in the outpatient supportive care center (SCC)
* History of use of non-medical opioid use (Screener and Opioid Assessment for Patients with Pain [SOAPP] >= 7+ and/or Cut Down, Annoyed, Guilty, and Eye opener questionnaire [CAGE] >= 2+)
* Physician-estimated prognosis of at least 12 months
* Age 18 or older
* Able to complete study assessments
* Willing to sign written informed consent
* Both human papillomavirus (HPV) and non-HPV patients will be included
* Patients currently receiving opioids for at least 1 week
* Able to read, write and speak English

Exclusion Criteria:

* Individual with clinically evident impaired cognition by Memorial Delirium Assessment Scale (MDAS) score of >= 13
* Employees of MD Anderson Cancer Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of non-medical opioid use (NMOU) behaviors | through study completion, an average of a year.
  Composite NMOU score is calculated by summing the number of times each behavior suggestive of NMOU is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org